CLINICAL TRIAL: NCT05579990
Title: Feasibility of a Meal Delivery Intervention for Postpartum Weight Management
Brief Title: Feasibility of Meal Delivery Postpartum
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Camille S Worthington, PhD, Primary Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB-300010155; U54MD000502 (NIH)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2025-08-05 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Postpartum Weight Retention; Obesity
Keywords: Postpartum; Weight management; Meal delivery
MeSH Terms: conditions — Gestational Weight Gain; Obesity

STUDY DESIGN:
Masking Description: All participants enrolled in the study will receive the meal delivery intervention, so blinding is not possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Meal Delivery (Experimental): Meal delivery intervention program designed to help low income postpartum women lose weight through weekly meal delivery and behavioral strategies.
  Interventions: Behavioral: Meal Delivery

INTERVENTIONS:
Behavioral: Meal Delivery — 10 home-delivered meals per week provided by a local meal delivery company supplemented by remote weekly behavioral support with study staff.

SUMMARY:
This study is being done to assess the feasibility and acceptability of a meal delivery intervention among low-income postpartum women with obesity.

DETAILED DESCRIPTION:
This is a single-group pilot study in which subjects will receive 10 home-delivered meals per week for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Medicaid eligible and/or have a household income at or below 185 percent of the federal poverty line
* 18 years of age or older
* Initiated prenatal care at a University of Alabama at Birmingham prenatal clinic
* Experienced a healthy singleton pregnancy
* 5-45 weeks postpartum at enrollment
* Body mass index >= 30 at enrollment
* Residing within the meal company's delivery radius
* Willing to consent

Exclusion Criteria:

* Self-reported major health condition (such as renal disease, cancer, or Type 1 or Type 2 diabetes)
* Current treatment for severe psychiatric disorder (such as schizophrenia)
* Self-reported diagnosis of anorexia or bulimia
* Current use of medication expected to significantly impact body weight
* Current substance abuse
* Participation in another dietary and/or weight management intervention postpartum
* Unable to understand and communicate in English
* Unwilling or unable to consume study meals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-09-27 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2025-09-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Camille S Worthington, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) that underlie the results reported in a publication will be made available upon request beginning 9 months and ending 36 months following article publication. The research team will keep a record of all individuals and/or research teams who request and receive a copy of the project data. Interested investigators will be asked to submit a document indicating the specific aims of the analyses, the analytic plan, available resources for completing the proposed project, proposed timeline, and goals (i.e., manuscripts, presentations, and/or grant applications). The PI and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after publication of results and ending 36 months following article publication.
Access Criteria: Access to IPD stripped of all HIPAA identifiers (except age) for this study can be requested by qualified researchers engaging in independent scientific research whose proposed research has received Institutional Review Board approval, and will be provided following review and approval of a research proposal and timeline, statistical analysis plan, and goals (e.g., manuscripts, presentations, grant applications). The Principal Investigator (PI) and research team will review these requests to determine whether the proposed analyses constitute an innovative and significant exploration of the data, whether the proposed team has sufficient resources to complete the request, and whether data will be adequately protected and managed. Based on institutional policies, execution of a Data Sharing Agreement may be required prior to sharing of IPD. IPD requests can be made to the PI at cschneid@uab.edu.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Not applicable as there was no randomization. All participants began receiving the meal delivery intervention after completing enrollment and baseline assessment measures.
Groups:
- Meal Delivery: Meal delivery intervention program designed to help low-income postpartum women lose weight through weekly meal delivery and behavioral strategies.
  Meal Delivery: 10 home-delivered meals per week for 8 weeks provided by a local meal delivery company supplemented by remote weekly behavioral support with study staff.
Period: Overall Study
Arm/Group | Meal Delivery
Started | 11
Completed | 8
Not Completed | 3
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Arm/Group | Meal Delivery
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.5 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 8
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Participant Overall Satisfaction with Diet [Mean (Standard Deviation); unit: score on a scale] — To assess satisfaction with the study intervention, the 28-item Diet Satisfaction Questionnaire (DSAT-28) was used in which participants respond to 28 statements using a 5-point Likert scale. Responses are averaged to produce an overall total diet satisfaction score ranging from 1-5. Higher scores represent greater satisfaction. The overall diet satisfaction score is designed to reflect satisfaction as it relates to following a weight-management diet.
  score on a scale | 2.95 (0.42)
Diet Satisfaction- Cost Factor [Mean (Standard Deviation); unit: score on a scale] — To assess satisfaction with the study intervention, the 28-item Diet Satisfaction Questionnaire was used in which participants respond to 28 statements using a 5-point Likert scale. Responses to 5-items related specifically to cost of the diet are averaged to produce a Cost Factor score ranging from 1-5. Higher scores represent greater satisfaction. The Cost Factor subscale score reflects financial cost of the diet.
  score on a scale | 2.87 (0.72)
Diet Satisfaction-Planning & Preparation Factor [Mean (Standard Deviation); unit: score on a scale] — To assess satisfaction with the study intervention, the 28-item Diet Satisfaction Questionnaire was used in which participants respond to 28 statements using a 5-point Likert scale. Responses to 5-items related specifically to meal planning and preparation are averaged to produce a Planning & Preparation Factor score ranging from 1-5. Higher scores represent greater satisfaction. The Planning & Preparation Factor score reflects the amount of time and effort spent in planning and preparing the diet.
  score on a scale | 3.44 (0.76)
Body Weight [Mean (Standard Deviation); unit: kilograms] — Body weight in kilograms measured at the baseline assessment.
  kilograms | 100.3 (15.4)
Food Security Score [Mean (Standard Deviation); unit: score on a scale] — Determined using the 18-item United States (US) Household Food Security Survey Module based on the previous 30 days. Adult food security scores range from 0 to 10, with lower values indicating greater food security.
  score on a scale | 1.5 (2.8)
Perceived Stress [Mean (Standard Deviation); unit: score on a scale] — Determined using the 10-item Perceived Stress Scale (PSS-10) based on the last month. PSS-10 scores range from 0 to 40, with higher scores representing higher levels of perceived stress.
  score on a scale | 12.7 (7.0)
Healthy Eating Self-Efficacy [Mean (Standard Deviation); unit: score on a scale] — Participants were asked to score 3 statements on a 5-point Likert scale ranging from 1=very sure to 5=very unsure (adapted from Lipsky LM et al. 2016). Responses are reverse coded and averaged, so higher scores reflect increasing self-efficacy.
  score on a scale | 3.8 (0.6)
Weight Control Self-Efficacy [Mean (Standard Deviation); unit: score on a scale] — Participants were asked to score 3 statements on a 5-point Likert scale ranging from 1=very sure to 5=very unsure (adapted from Lipsky LM et al. 2016). Responses are reverse coded and averaged, so higher scores reflect increasing self-efficacy.
  score on a scale | 3.0 (0.7)

OUTCOME MEASURES:

1. Primary Outcome: Self-Reported Proportion of Received Study Meals Consumed
Description: Proportion of received weekly study meals participants reported consuming each week collected via weekly electronic surveys in which participants will self-report the number of study meals a) they consumed, b) other household members consumed, or c) that were uneaten.
Time Frame: Collected weekly from intervention start (6-45 weeks postpartum) to follow-up (14-53 weeks postpartum)
Population: The total number of meals received were analyzed to determine the average proportion of provided study meals the participant reportd they ate, others in the household ate, and that were thrown away/frozen/uneaten per week. One participant did not receive meals for 2 weeks due to delivery errors, which is why the total units analyzed is 620.
Measure: Mean (Standard Deviation); unit: Proportion of Received Meals
Units Other Than Participants: Number of Meals Received
Arm/Group | Meal Delivery
Number analyzed (Participants) | 8
Number analyzed (Number of Meals Received) | 620
Proportion of Received Meals
  Proportion of Meals Participant Ate | 0.86 (0.25)
  Proportion of Meals Someone Else in Household Ate | 0.05 (0.11)
  Proportion of Meals thrown away/frozen/uneaten | 0.09 (0.24)

2. Secondary Outcome: Study Participation Rate
Description: Total number of eligible subjects who agreed to participate out of those who were screened.
Time Frame: baseline (5-45 weeks postpartum)
Population: The overall Number of Participants Analyzed (N=24) reflects the total number of participants who were screened, including those who may not have been eligible/consented into the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Delivery
Number analyzed (Participants) | 24
Participants | 11

3. Secondary Outcome: Participant Retention
Description: The number of enrolled participants who completed some or all follow-up assessment visit measurements.
Time Frame: baseline (5-45 weeks postpartum), follow-up (14-53 weeks postpartum)
Population: The overall number of participants analyzed (N=11) reflects the number of participants who enrolled in the study, including those who completed all of the 8-week follow-up assessment measurements, those who completed some (but not all) of the 8-week follow-up assessment measurements, and those that did not complete any of the 8-week follow-up assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Meal Delivery
Number analyzed (Participants) | 11
Participants
  Completed all follow-up measurements | 6
  Completed some (but not all) follow up measurements | 2

4. Secondary Outcome: Change in Participant Satisfaction With Diet
Description: To assess satisfaction with the study intervention, the 28-item Diet Satisfaction Questionnaire (DSAT-28) will be used in which participants respond to 28 statements using a 5-point Likert scale. Responses to all 28-items are averaged to produce a total diet satisfaction score (designed to reflect satisfaction as it relates to following a weight-management diet) ranging from 1-5. Subscale scores for Cost Factor (reflects financial cost of the diet) and Planning & Preparation Factor (reflects amount of time and effort spent in planning and preparing) will also be calculated and range from 1-5. For the overall diet satisfaction score and subscale scores, higher scores represent greater satisfaction. Changes in overall diet satisfaction, as well as changes in subscale scores for Cost Factor and Planning & Preparation Factor will be examined from baseline to follow-up.
Time Frame: baseline (5-45 weeks postpartum), follow-up (14-53 weeks postpartum)
Population: Change calculated as score at 8-week follow up minus score at baseline, with positive values indicating an increase in score (which reflects an increase in satisfaction) from baseline to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meal Delivery
Number analyzed (Participants) | 6
score on a scale
  Change in overall diet satisfaction score | 0.17 (0.5)
  Change in Cost Factor Score | 0.3 (0.8)
  Change in Planning & Preparation Factor Score | -0.2 (0.9)

5. Other Pre Specified Outcome: Change in Weight
Description: Body weight measured at baseline and follow-up will be used to calculate weight change.
Time Frame: baseline (5-45 weeks postpartum), follow-up (14-53 weeks postpartum)
Population: Change calculated as weight at 8-week follow up minus weight at baseline, with negative values indicating weight loss from baseline to follow up.
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Meal Delivery
Number analyzed (Participants) | 7
kilograms | -0.18 (4.77)

6. Other Pre Specified Outcome: Change in Food Security
Description: Determined using the 18-item United States (US) Household Food Security Survey Module based on the previous 30 days. Adult food security scores range from 0 to 10, with lower values indicating greater food security.
Time Frame: baseline (5-45 weeks postpartum), follow-up (14-53 weeks postpartum)
Population: Change calculated as food security score at 8-week follow up minus score at baseline, with negative values indicating an increase in food security from baseline to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meal Delivery
Number analyzed (Participants) | 6
score on a scale | -0.5 (0.8)

7. Other Pre Specified Outcome: Change in Perceived Stress
Description: Determined using the 10-item Perceived Stress Scale (PSS-10) based on the last month. PSS-10 scores range from 0 to 40, with higher scores representing higher levels of perceived stress.
Time Frame: baseline (5-45 weeks postpartum), follow-up (14-53 weeks postpartum)
Population: Change calculated as score at 8-week follow up minus score at baseline, with positive values indicating an increase in perceive stress score from baseline to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meal Delivery
Number analyzed (Participants) | 6
score on a scale | 1.8 (5.9)

8. Other Pre Specified Outcome: Change in Healthy Eating Self-Efficacy
Description: Participants will be asked to score 3 statements on a 5-point Likert scale ranging from 1=very sure to 5=very unsure (adapted from Lipsky LM et al. 2016). Responses are reverse coded and averaged, so higher scores reflect increasing self-efficacy.
Time Frame: baseline (5-45 weeks postpartum), follow-up (14-53 weeks postpartum)
Population: Change calculated as score at 8-week follow up minus score at baseline, with positive values indicating an increase in self-efficacy from baseline to follow up.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meal Delivery
Number analyzed (Participants) | 6
score on a scale | -0.6 (0.9)

9. Other Pre Specified Outcome: Change in Weight Control Self-Efficacy
Description: as for outcome 8
Time Frame: baseline (5-45 weeks postpartum), follow-up (14-53 weeks postpartum)
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Meal Delivery
Number analyzed (Participants) | 6
score on a scale | 0.38 (0.57)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected via weekly electronic surveys sent each week during the 8-week study meal delivery intervention period.
Description: Adverse event data were collected via weekly electronic surveys sent each week during the 8-week study meal delivery intervention period.
Arm/Group | Meal Delivery
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 1/11
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Meal Delivery (N=11)
Emesis (Gastrointestinal disorders) | 1 (1) — There was a single instance of a participant reporting one episode of emesis once during the intervention.
Diarrhea (Gastrointestinal disorders) | 1 (1) — There was a single instance of a participant reporting having diarrhea once during the intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2025-04-10): https://cdn.clinicaltrials.gov/large-docs/90/NCT05579990/Prot_SAP_ICF_000.pdf